CLINICAL TRIAL: NCT04495946
Title: Implementation and Effectiveness of Engagement and Collaborative Management to Proactively Advance Sepsis Survivorship: A Hybrid Effectiveness-Implementation Randomized Controlled Trial
Brief Title: Implementation and Effectiveness of Engagement and Collaborative Management to Proactively Advance Sepsis Survivorship
Acronym: ENCOMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00081729; R01NR018434 (NIH); Pro00036873 (Other: Atrium Health)
Record Dates: First submitted 2020-07-07; First posted 2020-08-03 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-05

CONDITIONS: Sepsis
Keywords: evidence based medicine; transition care; critical care; implementation science; pragmatic clinical trial
MeSH Terms: conditions — Sepsis | interventions — Salvage Therapy

STUDY DESIGN:
Intervention Model Description: Pragmatic, stepped-wedge cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sepsis Transition and Recovery (STAR) Program (Experimental): Virtual sepsis navigation delivered across the peri-hospital discharge interval
  Interventions: Behavioral: Sepsis Transition and Recovery (STAR) program
- Usual Care (Active Comparator): Standard of care received through Atrium Health facilities for patients hospitalized with sepsis. Aspects of usual care will be determined by treating clinicians independent of trial assignment.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Sepsis Transition and Recovery (STAR) program — In the STAR program intervention, a centrally located nurse navigator facilitates the application of four evidence-based core components of post-sepsis care (i.e., review of medications, new impairments, comorbidities, and palliative care) to patients prior to and during the 90 days after hospital discharge. The STAR navigator will provide telephone and EHR-based support within the hospitalization and to patients across all discharge settings with remote monitoring at specified intervals following hospital discharge. Patients will continue to receive STAR directed services for 90 days following their discharge and then will be transitioned back to the next appropriate care location.
  Arms: Sepsis Transition and Recovery (STAR) Program
Behavioral: Usual care — Hospitals and their patients will not have access to the STAR program. Patients will continue to receive usual care throughout their stay and discharge, consisting of: patient education and follow-up instructions at discharge, which are not specific to sepsis; routine recommendations for follow-up visits with primary care providers; arrangements for home health services or care management follow-up based on each patient's needs but not specifically tailored to the sepsis population; discharge to post-acute setting with no sepsis-specific follow-up. All aspects of usual care will be determined by treating clinicians independent of trial assignment.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate if implementation of the Sepsis Transition and Recovery (STAR) program within a large healthcare system will improve outcomes for high-risk patients with suspected sepsis, while concurrently examining contextual factors related to STAR program delivery within routine care to generate knowledge of best practices for implementation and dissemination of post sepsis transitions of care. To address persistent morbidity and mortality for sepsis survivors, Atrium Health developed the Sepsis Treatment and Recovery (STAR) program which uses a nurse navigator to deliver a bundle of best-practice care elements for the delivery of longitudinal post-sepsis care for up to 90 days. These care elements are directed towards the specific challenges and sequelae following a sepsis hospitalization and include: 1) identification and treatment of new physical, mental, and cognitive deficits; 2) review and adjustment of medications; 3) surveillance of treatable conditions that commonly lead to poor outcomes including chronic conditions that may de-stabilize during sepsis and recovery; and 4) focus on palliative care when appropriate. ENCOMPASS (Engagement and Collaborative Management to Proactively Advance Sepsis Survivorship) is an effectiveness-implementation hybrid type I trial, with the evaluation designed as a two-arm, pragmatic, stepped-wedge cluster randomized controlled trial conducted at eight regional hospitals in which each participating hospital begins in a usual care control phase and transitions to the STAR program intervention in a randomly assigned sequence. Patients are allocated to receive the treatment condition (i.e., usual care or STAR) assigned to their admission hospital at time of enrollment. ENCOMPASS will test the hypothesis that patients who receive care through the STAR program will have reduced mortality and hospital readmission assessed 90 days post index hospital discharge compared to patients who receive usual care.

DETAILED DESCRIPTION:
BACKGROUND

Sepsis is a common and life-threatening condition defined by organ dysfunction due to a dysregulated response to infection (Fleischmann, 2016). Aggressive early sepsis identification and treatment initiatives have decreased hospital mortality for patients with sepsis (Rhodes, 2017; Kaukonen, 2014). However, sepsis survivors continue to face challenges after the acute illness episode, experiencing new functional, cognitive, and psychological deficits, and high rates of hospital readmission and mortality in the 90-days after hospital discharge (Iwashyna, 2010; Borges, 2015; Annane, 2015; Prescott, 2015; Mayr, 2017). To address persistent morbidity and mortality for sepsis survivors, Atrium Health developed the Sepsis Treatment and Recovery (STAR) program which uses a nurse navigator to deliver a bundle of best-practice care elements for the delivery of longitudinal post-sepsis care for up to 90 days. These care elements are directed towards the specific challenges and sequelae following a sepsis hospitalization and include: 1) identification and treatment of new physical, mental, and cognitive deficits; 2) review and adjustment of medications; 3) surveillance of treatable conditions that commonly lead to poor outcomes including chronic conditions that may destabilize during sepsis and recovery; and 4) focus on palliative care when appropriate (Prescott, 2018) These care elements have good face-validity and have shown to be associated with improved outcomes for sepsis survivors in observational data (Taylor, 2020). However, they are not widely applied in real-world settings for this vulnerable population, likely hindered by a gap in understanding key contextual factors underlying how to best integrate this bundle of care elements into the complex and fragmented post-discharge setting (Brownson, 2012; Bodenheimer, 2008; Coleman, 2004; Kim, 2013)

RATIONALE

In randomized controlled trials (RCTs), successfully implemented care transition programs using nurse navigators have been shown to reduce hospital readmission and costs. To better enhance transitions of care for the highest risk, complex patients with suspected sepsis, the investigators propose extending this evidence using a nurse-facilitated care transition program for patients in the post-sepsis transition period to improve the implementation of recommended care practices and bridge care gaps. This approach, called the Sepsis Transition and Recovery (STAR) program, is the next step in the progression of the investigator team's work on improving discharge transitions and sepsis processes of care. A key aspect of this initiative includes the ability to identify sepsis survivors at the greatest risk for poor outcomes. For example, one-quarter of sepsis survivors account for three-quarters of hospital readmission and costs, indicating that identifying high-risk sepsis patients for targeted facilitation of best-practice care could efficiently impact quality and cost.

The STAR program uses near real-time risk modeling to identify high-risk patients and a centrally located nurse, virtually connected to participating hospitals, to coordinate the application of evidence-based recommendations for post-sepsis care, overcome barriers to recommended care, and bridge gaps in service that can serve as points of failure for complex patients. During hospitalization, high-risk patients enter into a transition pathway integrated within Atrium Health Hospital Medicine's Transition Services program and includes the following core components: i) Introduction to STAR process prior to discharge (confirm provider consults e.g., PT, ID, palliative); ii) Disease-specific education and discharge "playbook"; iii) Virtual hospital follow-up evaluation within 48 hours including medication reconciliation; iv) Second, post-acute virtual follow-up within 72-96 hours (symptom monitoring, confirm provider follow-up); v) Weekly contact with STAR team; vi) Referral to provider follow-up (e.g., primary care provider, transition clinic) as appropriate; vii) Coordinated transition to the next appropriate care location after 90 days from time of discharge. The STAR navigator also meets weekly with the Medical Director of the Atrium Health Transition Services program who provides additional clinical oversight of ongoing cases.

The ENCOMPASS (Engagement and Collaborative Management to Proactively Advance Sepsis Survivorship) evaluation will examine if implementation of the STAR program within a large healthcare system will improve outcomes for high-risk sepsis patients. This cluster randomized program evaluation is designed to be a seamless part of routine care in a real-world setting to generate knowledge of best practices for implementation and dissemination of post-sepsis transitions of care.

INVESTIGATIONAL PLAN

Overall Study Design ENCOMPASS is an effectiveness-implementation hybrid type I trial. The evaluation component is designed as a two-arm, pragmatic, stepped-wedge cluster randomized controlled trial conducted at eight regional hospitals in which each participating hospital begins in a usual care control phase and transitions to the STAR program intervention in a randomly assigned sequence, with one of eight hospitals assigned to transition at each four-month interval (i.e., step). During the time that a hospital is allocated to usual care, all eligible patients will receive usual care. Once a hospital has been allocated to the STAR arm, all eligible patients will receive STAR during their index hospitalization and extending through 90 days from discharge or date of death. The ENCOMPASS trial will compare the effectiveness of the Sepsis Transition And Recovery (STAR) program versus usual care on post-sepsis care and patient outcomes. The STAR program is informed by existing evidence and designed using the Chronic Care Model to increase best-practice adherence and care coordination, resulting in improved transitions between hospitals and post-acute care during sepsis recovery.

ENCOMPASS will test the STAR program intervention within the course of providing usual care among a large and diverse population of post-sepsis patients admitted to eight hospitals within Atrium Health, one of the largest, vertically integrated health systems in the US. The eight acute care hospitals participating in this study use the same EHR, which connects across all points of care, including outpatient practices, urgent care locations, emergency departments and hospitals. Consistent with the pragmatic study design concept, eligibility criteria are broad, the sample size is large and diverse, and study procedures are embedded into the context of routine care. To be objective in patient selection and allow for program evaluation, a data driven approach will be used to identify patients as eligible for program referral. Each weekday morning actively admitted patients at eight study hospitals will be identified from the electronic health record and Enterprise Data Warehouse and output into daily eligibility lists based on the study's inclusion/exclusion criteria. Primary analyses will be conducted using an intent-to-treat approach such that all eligible patients will be included. Planned enrollment is 4032 patients and STAR program follow-up will be completed 90 days after hospital discharge. Outcomes data will be tracked for 90 days and captured from routinely collected data from the Atrium Health Enterprise Data Warehouse. Given this evaluation protocol relies on using evidence-based interventions, only utilizes data collected as part of routine care, and is minimal risk to patients, the institutional review board granted the request for waiver of informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age upon admission
2. Suspected infection

   1. Oral/parenteral antibiotic or bacterial culture order within 24 hours of emergency department presentation; and
   2. Evidence of systemic inflammatory response (i.e., at least two abnormal of temperature; heart rate; respiratory rate; and WBC count or bands)
3. Evidence of organ dysfunction (i.e., at least two points on either Quick Sepsis-related Organ Failure Assessment or Sepsis-related Organ Failure Assessment risk tools)
4. Deemed as high risk for 90-day readmission using risk-scoring models
5. Not discharged at the time of patient list generation

Exclusion Criteria:

1. Patients with a change in code status (i.e., do not resuscitate, do not intubate) within 24 hours after infection onset due to presumed limitation of aggressive treatment
2. Patients who reside > 2.5 hours drive time from the treating hospital
3. Patients actively enrolled in a different care management program at time of admission
4. Patient has been randomized previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3894 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kowalkowski, PhD, Principal Investigator — Wake Forest University Health Sciences; Stephanie P Taylor, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Borges RC, Carvalho CR, Colombo AS, da Silva Borges MP, Soriano FG. Physical activity, muscle strength, and exercise capacity 3 months after severe sepsis and septic shock. Intensive Care Med. 2015 Aug;41(8):1433-44. doi: 10.1007/s00134-015-3914-y. Epub 2015 Jun 25. PMID 26109398
- [Background] Annane D, Sharshar T. Cognitive decline after sepsis. Lancet Respir Med. 2015 Jan;3(1):61-9. doi: 10.1016/S2213-2600(14)70246-2. Epub 2014 Nov 28. PMID 25434614
- [Background] Prescott HC, Langa KM, Iwashyna TJ. Readmission diagnoses after hospitalization for severe sepsis and other acute medical conditions. JAMA. 2015 Mar 10;313(10):1055-7. doi: 10.1001/jama.2015.1410. No abstract available. PMID 25756444
- [Background] Mayr FB, Talisa VB, Balakumar V, Chang CH, Fine M, Yende S. Proportion and Cost of Unplanned 30-Day Readmissions After Sepsis Compared With Other Medical Conditions. JAMA. 2017 Feb 7;317(5):530-531. doi: 10.1001/jama.2016.20468. No abstract available. PMID 28114505
- [Background] Prescott HC, Angus DC. Enhancing Recovery From Sepsis: A Review. JAMA. 2018 Jan 2;319(1):62-75. doi: 10.1001/jama.2017.17687. PMID 29297082
- [Background] Taylor SP, Chou SH, Sierra MF, Shuman TP, McWilliams AD, Taylor BT, Russo M, Evans SL, Rossman W, Murphy S, Cunningham K, Kowalkowski MA. Association between Adherence to Recommended Care and Outcomes for Adult Survivors of Sepsis. Ann Am Thorac Soc. 2020 Jan;17(1):89-97. doi: 10.1513/AnnalsATS.201907-514OC. PMID 31644304
- [Background] Brownson RC, Allen P, Duggan K, Stamatakis KA, Erwin PC. Fostering more-effective public health by identifying administrative evidence-based practices: a review of the literature. Am J Prev Med. 2012 Sep;43(3):309-19. doi: 10.1016/j.amepre.2012.06.006. PMID 22898125
- [Background] Bodenheimer T. Coordinating care--a perilous journey through the health care system. N Engl J Med. 2008 Mar 6;358(10):1064-71. doi: 10.1056/NEJMhpr0706165. No abstract available. PMID 18322289
- [Background] Coleman EA, Berenson RA. Lost in transition: challenges and opportunities for improving the quality of transitional care. Ann Intern Med. 2004 Oct 5;141(7):533-6. doi: 10.7326/0003-4819-141-7-200410050-00009. PMID 15466770
- [Background] Kim CS, Flanders SA. In the Clinic. Transitions of care. Ann Intern Med. 2013 Mar 5;158(5 Pt 1):ITC3-1. doi: 10.7326/0003-4819-158-5-201303050-01003. No abstract available. PMID 23460071
- [Derived] Taylor SP, Eaton T, Rios A, Boyd D, Tapp H, McWilliams A, Chou SH, Halpern S, Angus DC, McCurdy L, Ganesan A, Nguyen H, Connor CD, Kowalkowski M. Proactive Telehealth-Based Sepsis Transition and Recovery Support, Hospital Readmission, and Mortality: A Randomized Clinical Trial. JAMA Intern Med. 2025 Oct 1;185(10):1238-1246. doi: 10.1001/jamainternmed.2025.3699. PMID 40788609
- [Derived] Eaton TA, Kowalkowski M, Burns R, Tapp H, O'Hare K, Taylor SP. Pre-implementation planning for a sepsis intervention in a large learning health system: a qualitative study. BMC Health Serv Res. 2024 Aug 28;24(1):996. doi: 10.1186/s12913-024-11344-x. PMID 39192331
- [Derived] Kowalkowski M, Eaton T, McWilliams A, Tapp H, Rios A, Murphy S, Burns R, Gutnik B, O'Hare K, McCurdy L, Dulin M, Blanchette C, Chou SH, Halpern S, Angus DC, Taylor SP. Protocol for a two-arm pragmatic stepped-wedge hybrid effectiveness-implementation trial evaluating Engagement and Collaborative Management to Proactively Advance Sepsis Survivorship (ENCOMPASS). BMC Health Serv Res. 2021 Jun 2;21(1):544. doi: 10.1186/s12913-021-06521-1. PMID 34078374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a 36-month stepped-wedge cluster randomized trial. Each hospital begins enrolling patients under usual care and transitions to enrolling patients in STAR program one hospital at a time in a randomly determined sequence every 4 months. The randomization sequence was concealed to all hospitals until 1 month before each individual hospital transitioned to receive the STAR program. The trial was conducted at 7 hospitals in the Atrium Health system and one additional outside hospital.
Pre-assignment Details: The outside hospital affiliated with a different health system withdrew from the trial after randomization but prior to receiving the intervention.
  The number of participants to start a Period is not equal to the number who completed the previous Period since this is a pragmatic trial with cross-sectional sampling of eligible patients in each step at each participating study site.
Groups:
- Sequence 1: 4m Usual Care Then 32m STAR (Hospital A); Sequence 2: 8m Usual Care Then 28m STAR (Hospital B); Sequence 3: 12m Usual Care Then 24m STAR (Hospital C); Sequence 4: 16m Usual Care Then 20m STAR (Hospital D); Sequence 5: 20m Usual Care Then 16m STAR (Hospital E); Sequence 6: 24m Usual Care Then 12m STAR (Hospital F); Sequence 7: 28m Usual Care Then 8m STAR (Hospital G); Sequence 8: 32m Usual Care Then 4m STAR (Hospital H): During Usual Care, hospitals and their patients will not have access to the STAR program. Patients will continue to receive usual care throughout their stay and discharge, consisting of: patient education and follow-up instructions at discharge, which are not specific to sepsis; routine recommendations for follow-up visits with primary care providers; arrangements for home health services or care management follow-up based on each patient's needs but not specifically tailored to the sepsis population; discharge to post-acute setting with no sepsis-specific follow-up. All aspects of usual care will be determined by treating clinicians independent of trial assignment.
  During the STAR program intervention, a centrally located nurse navigator facilitates the application of four evidence-based core components of post-sepsis care (i.e., review of medications, new impairments, comorbidities, and palliative care) to patients prior to and during the 90 days after hospital discharge. The STAR navigator will provide telephone and EHR-based support within the hospitalization and to patients across all discharge settings with remote monitoring at specified intervals following hospital discharge. Patients will continue to receive STAR directed services for 90 days following their discharge and then will be transitioned back to the next appropriate care location.
Period: Step 1: 4m (July 2020-Oct 2020)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 98 | 8 | 48 | 79 | 88 | 37 | 44 | 66
Completed | 98 | 8 | 48 | 79 | 88 | 37 | 44 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 66
Period: Step 2: 4m (Nov 2020-Feb 2021)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 106 | 6 | 49 | 51 | 90 | 45 | 43 | 48
Completed | 106 | 6 | 49 | 51 | 90 | 45 | 43 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 48
Period: Step 3: 4m (Mar 2021-Jun 2021)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 108 | 6 | 45 | 67 | 94 | 41 | 27 | 60
Completed | 108 | 6 | 45 | 67 | 94 | 41 | 27 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 60
Period: Step 4: 4m (Jul 2021-Oct 2021)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 90 | 9 | 49 | 66 | 84 | 36 | 37 | 52
Completed | 90 | 9 | 49 | 66 | 84 | 36 | 37 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 52
Period: Step 5: 4m (Nov 2021-Feb 2022)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 92 | 9 | 57 | 62 | 75 | 44 | 39 | 63
Completed | 92 | 9 | 57 | 62 | 75 | 44 | 39 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63
Period: Step 6: 4m (Mar 2022-Jun 2022)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 87 | 6 | 33 | 61 | 51 | 34 | 18 | 45
Completed | 87 | 6 | 33 | 61 | 51 | 34 | 18 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45
Period: Step 7: 4m (Jul 2022-Oct 2022)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 114 | 9 | 36 | 81 | 88 | 44 | 33 | 12
Completed | 114 | 9 | 36 | 81 | 88 | 44 | 33 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
Period: Step 8: 4m (Nov 2022-Feb 2023)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 135 | 7 | 41 | 93 | 111 | 41 | 52 | 0
Completed | 135 | 7 | 41 | 93 | 111 | 41 | 52 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 9: 4m (Mar 2023-Jun 2023)
Arm/Group | Sequence 1: 4m Usual Care Then 32m STAR (Hospital A) | Sequence 2: 8m Usual Care Then 28m STAR (Hospital B) | Sequence 3: 12m Usual Care Then 24m STAR (Hospital C) | Sequence 4: 16m Usual Care Then 20m STAR (Hospital D) | Sequence 5: 20m Usual Care Then 16m STAR (Hospital E) | Sequence 6: 24m Usual Care Then 12m STAR (Hospital F) | Sequence 7: 28m Usual Care Then 8m STAR (Hospital G) | Sequence 8: 32m Usual Care Then 4m STAR (Hospital H)
Started | 141 | 3 | 41 | 78 | 110 | 31 | 39 | 0
Completed | 141 | 3 | 41 | 78 | 110 | 31 | 39 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care | Total
Number analyzed (Participants) | 2122 | 1426 | 3548
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age at hospital admission, in years
  years | 65.65 (15.07) | 65.44 (15.37) | 65.56 (15.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1056 | 787 | 1843
  Male | 1066 | 639 | 1705
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 4 | 12
  Asian | 26 | 4 | 30
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 499 | 368 | 867
  White | 1537 | 1031 | 2568
  More than one race | 12 | 10 | 22
  Unknown or Not Reported | 39 | 9 | 48
Sequential Organ Failure Assessment (SOFA) score [Mean (Standard Deviation); unit: units on a scale] — Mean SOFA score at hospital admission, with a score range from 0 to 24 points (higher is worse)
  units on a scale | 4.635 (2.521) | 4.647 (2.378) | 4.637 (2.464)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality and Hospital Readmission Rate
Description: Combined death or unplanned hospital readmission due to any cause, assessed 90 days after the index hospital discharge
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 1023 | 684

2. Secondary Outcome: Number of Days Alive and Outside the Hospital
Description: The total days alive without inpatient, observation, and emergency department care utilization beginning with the day of index hospital admission and ending 90 days after discharge or on the date of death if prior to 90 days.
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Days | 72.2 [71.9 to 72.6] | 71.9 [70.5 to 73.3]

3. Secondary Outcome: All-cause Mortality Rate
Description: Patients with date of death prior to 90 days post discharge documented in the electronic health record or in linked national death records
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 367 | 292

4. Secondary Outcome: All-cause Hospital Readmission Rate
Description: Any hospital readmission, including both inpatient and observation status hospitalizations, assessed 90 days post index hospital discharge.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 763 | 478

5. Secondary Outcome: Number of Outpatient Provider Visits
Description: Number of outpatient provider visits assessed 90 days post index hospital discharge
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: count of visits
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
count of visits | 3.0 [2.8 to 3.2] | 3.6 [3.4 to 3.9]

6. Secondary Outcome: Number of Emergency Department Visits
Description: Number of emergency department visits assessed 90 days post index hospital discharge
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: count of visits
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
count of visits | 0.50 [0.44 to 0.55] | 0.46 [0.40 to 0.51]

7. Secondary Outcome: Cause-specific Hospital Readmission Rate
Description: Any hospital readmission due to sepsis or other infection conditions assessed 90 days post index hospital discharge
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 370 | 222

8. Secondary Outcome: Inpatient Functional Assessment or Physical Therapy Consult
Description: Documented inpatient functional assessment or physical therapy consult completed and captured from electronic health records
Time Frame: Index hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 1768 | 1196

9. Secondary Outcome: Inpatient Mental Health Assessment
Description: Documented inpatient mental health assessment completed and captured from electronic health records
Time Frame: Index hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 2048 | 1385

10. Secondary Outcome: Count of Participants With Support Service Referrals
Description: Outpatient rehabilitation or physical, occupational, or speech therapy during follow-up
Time Frame: 90 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 594 | 374

11. Secondary Outcome: Early Outpatient Provider Follow up
Description: The completion of hospital follow-up visit with an outpatient provider within 7 days of hospital discharge captured from electronic health records
Time Frame: 7 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 468 | 348

12. Secondary Outcome: Outpatient Medication Reconciliation
Description: Completion of medication reconciliation in the electronic health record during the 90 days post hospital discharge
Time Frame: 90 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 1590 | 866

13. Secondary Outcome: Palliative Care Consultation
Description: Documented completion of palliative care consult captured from electronic health records.
Time Frame: Index hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 430 | 234

14. Secondary Outcome: Completed Care Preferences
Description: Documented completion of patient care preferences form captured from electronic health records
Time Frame: Index hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 526 | 309

15. Secondary Outcome: Discharge to Hospice Care
Description: Discharge disposition of hospice care from initial sepsis hospitalization captured from electronic health records
Time Frame: Index hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants | 97 | 69

16. Secondary Outcome: Place of Death
Description: In-hospital, hospice, and home or other location of death captured from electronic health records
Time Frame: 90 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
Number analyzed (Participants) | 2122 | 1426
Participants
  In hospital deaths | 204 | 150
  Hospice deaths | 69 | 67
  Home or other deaths | 94 | 75

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow up, up to 90 days after hospital discharge
Arm/Group | Sepsis Transition and Recovery (STAR) Program | Usual Care
All-Cause Mortality (participants affected / at risk) | 367/2122 | 292/1426
Serious Adverse Events (participants affected / at risk) | 763/2122 | 478/1426
Other Adverse Events (participants affected / at risk) | 0/2122 | 0/1426
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sepsis Transition and Recovery (STAR) Program (N=2122) | Usual Care (N=1426)
Disease complications experienced during 90 day follow up that required rehospitalization (General disorders) | 763 | 478

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT04495946/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04495946/ICF_000.pdf